CLINICAL TRIAL: NCT04401657
Title: Relationship Between Fractional Flow Reserve and Inducible Myocardial Ischemia During Adenosine Stress Testing
Brief Title: FFR and Inducible Myocardial Ischemia During Adenosine Stress Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, CHEOL WHAN LEE, M.D., Ph.D, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FFR_Ischemia
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Stenosis
Keywords: Coronary artery disease; Myocardial ischemia; Fractional flow reserve
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FFR Measurement (Experimental): Myocardia ischemia evaluation during adenosine stress testing
  Interventions: Diagnostic Test: Fractional flow reserve with adenosine stress testing

INTERVENTIONS:
Diagnostic Test: Fractional flow reserve with adenosine stress testing — ECG, FFR, and two-dimensional echocardiographic monitoring will be continued before, during and after adenosine infusion.

SUMMARY:
This is a prospective, single center study involving 150 patients with stable coronary artery disease undergoing coronary angiography for chest pain evaluation. The relationship between FFR values and inducible myocardial ischemia at the time of definite ischemia during adenosine stress testing will be investigated.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) is commonly used to search for ischemia-producing lesions during percutaneous coronary intervention (PCI), and its assessment becomes an integral part to guide PCI when objective evidences of inducible myocardial ischemia are not available. A transient imbalance between oxygen supply and demand leads to the ischemic cascade, which are typically accompanied by regional wall motion abnormalities or electrocardiographic changes as objective evidences of inducible myocardial ischemia.

FFR is a pressure-derived surrogate of coronary flow limitation defined as the ratio of distal coronary pressure to aortic pressure during maximal hyperemia. FFR has been indirectly validated against noninvasive stress tests, and large outcome trials support the benefit of FFR-guided PCI strategy. However, FFR is not a direct measurement of coronary flow, and myocardial ischemia depends on coronary flow rather than pressure. In fact, an experimental model shows that myocardial function can be maintained without evidences of myocardial ischemia despite low FFR. Furthermore, FFR did not predict improvement in symptoms or exercise performance after PCI, challenging the current threshold of FFR for discriminating ischemia-producing lesions.

The clinical benefit of FFR-guided PCI is certainly related to relief of inducible myocardial ischemia. However, there is little information to examine a direct link between FFR values and documented inducible ischemia at the time of FFR measurement. Therefore, the investigators investigate the relationship between FFR values and inducible myocardial ischemia at the time of definite ischemia during adenosine stress testing.

A 12-lead ECG recordings, FFR, and two-dimensional echocardiographic monitoring will be continued before, during and after adenosine infusion. When new regional wall motion abnormalities in echocardiography develop, adenosine infusion is ended and echocardiographic monitoring will be continued until left ventricular wall motion returns to normal. Apical (two-chamber, four-chamber and five chamber views) and parasternal long-axis and short-axis views will be recorded for offline analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* Patients undergoing coronary angiography
* Moderate to severe stenosis (diameter stenosis equal or more than 50 percent by visual examination) in one major epicardial coronary artery
* Normal left ventricular function without regional wall motion abnormality

Exclusion Criteria:

* Contraindications to adenosine stress test*
* ECG abnormalities (bundle branch block, LVH with strain, pacing rhythm, WPW)
* History of previous myocardial infarction
* Significant multi-vessel coronary artery disease (diameter stenosis equal or more than 50%)
* Hypertrophic cardiomyopathy
* Significant valvular heart disease
* Bronchial asthma or chronic obstructive lung disease
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* Current treatment for the active cancer
* Expected life expectancy < 1 year
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Definite myocardial ischemia | during adenosine stress testing
  Echocardiographic wall motion score index score by 17-segment model or ST segment elevation/depression by 12-lead ECG during adenosine stress testing

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Whan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No